CLINICAL TRIAL: NCT01377844
Title: Efficacy and Safety of EGT0001442 Compared With Placebo in Patients With Type 2 Diabetes Mellitus Inadequately Controlled by Diet and Exercise and up to One Oral Anti-diabetes Agent
Brief Title: Efficacy and Safety of EGT0001442 in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Theracos (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: THR-1442-C-418
Record Dates: First submitted 2011-06-13; First posted 2011-06-21 (Estimated); Results first posted 2021-06-16 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — bexagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EGT0001442 (Experimental): EGT0001442 capsule, 20 mg, daily, 96 weeks
  Interventions: Drug: EGT0001442
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EGT0001442
  Other Names: Bexagliflozin
  Arms: EGT0001442
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the efficacy of EGT0001442 in lowering glycosylated Hemoglobin (HbA1c, A laboratory test to diagnose three months average of blood sugar)levels at 24th week from baseline, when compared to placebo group(no diabetic medication given). The secondary aim of the study is to evaluate the efficacy of EGT0001442 in lowering fasting blood glucose at the weeks 2 and 24 and comparing the results with placebo group. This study assess the efficacy of EGT0001442 based on the proportion of subjects who reach the American Diabetes Association (ADA) target of HbA1c of < 7% in EGT0001442 group and comparison with placebo. The study also evaluates the effect of EGT0001442 on systolic, diastolic pressures, body weight and compare with the respective placebo groups.This study also assess the change from baseline in HbA1c overtime, from week 1 to week 96. Finally, to assess the safety of EGT0001442 in the Type 2 Diabetic patients (adult/maturity onset).

DETAILED DESCRIPTION:
EGT0001442 is a compound that may inhibit the effect of other compounds in the body known as sugar transporters. The use of EGT0001442 may enhance the elimination of glucose from the blood by increasing the amount of urine produced. Hence the blood glucose levels are significantly decreased and the efficacy of EGT001442 can be established by assessing the three months average blood glucose levels (HbA1c). Due to the increased urinary output, the effect of EGT001442 on blood pressure levels are also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥18 years old
* Diagnosed with type 2 diabetes
* Body mass index (BMI) ≤ 45 kg/m2
* HbA1c between 7 and 10% (inclusive) at screening
* FPG <250 mg/dL at screening for subjects not treated with oral anti-diabetic therapies or FPG <240 mg/dL at screening for subjects treated with anti-diabetic therapies
* Diabetes currently treated with diet and exercise only or diet and exercise along with one approved oral anti-diabetic agent
* If taking anti-diabetic medication, dose and regimen must be stable for past 3 months
* If taking anti-hypertensive medication, dose and regimen must be stable for past 3 months
* If taking lipid modifying therapy, dose and regimen must be stable for past 3 months
* Blood glucose <250 mg/dL based on finger stick blood glucose for all subjects at randomization

Exclusion Criteria:

* Hemoglobinopathy that affects HbA1c measurement
* Current use of injected therapy for treatment of diabetes (insulin or GLP-1 receptor based therapy)
* Genitourinary tract infection within 6 weeks of screening
* Greater than 2 episodes of genitourinary tract infection in the past year
* History of kidney stones, bladder malfunction or other significant risk factor for urinary tract infections
* eGFR, as calculated by the modification of diet in renal disease study equation (MDRD), < 50 mL/min/1.73 m2
* Abnormal tests of liver function ALT, AST or bilirubin ≥ 3x ULN
* Diagnosis of retinopathy or significant nephropathy (eGFR < 50 mL/min/1.73 m2
* Uncontrolled hypertension (systolic blood pressure >160 or diastolic blood pressure >95)
* Not willing to use effective birth control, if female with child-bearing potential
* Life expectancy < 2 years
* New York Heart Association (NYHA) Class 4 heart failure
* Sera positive of HCV, HIV, or positive on drug screen
* Currently participating in another interventional trial
* Previous treatment with EGT0001442 or EGT0001474
* Not able to comply with the study scheduled visits

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2011-12; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mason W Freeman, M.D., Study Director — Massachusetts General Hospital
Locations (11):
- United States (11):
  - Site 5, Buena Park, California
  - Site 4, Los Angeles, California
  - Site 3, Santa Ana, California
  - Site 1, Hialeah, Florida
  - Site 9, Berlin, New Jersey
  - Site 7, Cary, North Carolina
  - Site 6, Marion, Ohio
  - Site 8, Munroe Falls, Ohio
  - Site 2, Portland, Oregon
  - Site 11, North Richland Hills, Texas
  - Site 7, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Diabetes Association. Standards of medical care in diabetes--2011. Diabetes Care. 2011 Jan;34 Suppl 1(Suppl 1):S11-61. doi: 10.2337/dc11-S011. No abstract available. PMID 21193625
- [Background] Ehrenkranz JR, Lewis NG, Kahn CR, Roth J. Phlorizin: a review. Diabetes Metab Res Rev. 2005 Jan-Feb;21(1):31-8. doi: 10.1002/dmrr.532. PMID 15624123
- [Background] Ferrannini E, Ramos SJ, Salsali A, Tang W, List JF. Dapagliflozin monotherapy in type 2 diabetic patients with inadequate glycemic control by diet and exercise: a randomized, double-blind, placebo-controlled, phase 3 trial. Diabetes Care. 2010 Oct;33(10):2217-24. doi: 10.2337/dc10-0612. Epub 2010 Jun 21. PMID 20566676
- [Background] Han S, Hagan DL, Taylor JR, Xin L, Meng W, Biller SA, Wetterau JR, Washburn WN, Whaley JM. Dapagliflozin, a selective SGLT2 inhibitor, improves glucose homeostasis in normal and diabetic rats. Diabetes. 2008 Jun;57(6):1723-9. doi: 10.2337/db07-1472. Epub 2008 Mar 20. PMID 18356408
- [Background] Komoroski B, Vachharajani N, Boulton D, Kornhauser D, Geraldes M, Li L, Pfister M. Dapagliflozin, a novel SGLT2 inhibitor, induces dose-dependent glucosuria in healthy subjects. Clin Pharmacol Ther. 2009 May;85(5):520-6. doi: 10.1038/clpt.2008.251. Epub 2009 Jan 7. PMID 19129748
- [Background] Komoroski B, Vachharajani N, Feng Y, Li L, Kornhauser D, Pfister M. Dapagliflozin, a novel, selective SGLT2 inhibitor, improved glycemic control over 2 weeks in patients with type 2 diabetes mellitus. Clin Pharmacol Ther. 2009 May;85(5):513-9. doi: 10.1038/clpt.2008.250. Epub 2009 Jan 7. PMID 19129749
- [Background] Neumiller JJ, White JR Jr, Campbell RK. Sodium-glucose co-transport inhibitors: progress and therapeutic potential in type 2 diabetes mellitus. Drugs. 2010 Mar 5;70(4):377-85. doi: 10.2165/11318680-000000000-00000. PMID 20205482
- [Background] Santer R, Kinner M, Lassen CL, Schneppenheim R, Eggert P, Bald M, Brodehl J, Daschner M, Ehrich JH, Kemper M, Li Volti S, Neuhaus T, Skovby F, Swift PG, Schaub J, Klaerke D. Molecular analysis of the SGLT2 gene in patients with renal glucosuria. J Am Soc Nephrol. 2003 Nov;14(11):2873-82. doi: 10.1097/01.asn.0000092790.89332.d2. PMID 14569097
- [Background] Sicree, R., Shaw, J., and Zimmet, P. (2010). The Global Burden - Diabetes and Impaired Glucose Tolerance (Baker IDI Heart and Diabetes Institute).
- [Background] van den Heuvel LP, Assink K, Willemsen M, Monnens L. Autosomal recessive renal glucosuria attributable to a mutation in the sodium glucose cotransporter (SGLT2). Hum Genet. 2002 Dec;111(6):544-7. doi: 10.1007/s00439-002-0820-5. Epub 2002 Sep 27. PMID 12436245

RESULTS

PARTICIPANT FLOW:
Groups:
- EGT0001442: EGT0001442 capsule, 20 mg, orally once daily
- Placebo: Placebo capsule, orally once daily
Period: Overall Study
Arm/Group | EGT0001442 | Placebo
Started | 145 | 143
Safety Population (Two subjects did not meet the eligibility criteria and were not dosed. They were excluded from the safety population.) | 145 | 141
Completed | 109 | 108
Not Completed | 36 | 35
Not completed — Withdrawal by Subject | 25 | 28
Not completed — Protocol Violation | 2 | 3
Not completed — Adverse Event | 3 | 0
Not completed — Physician Decision | 6 | 3
Not completed — Study terminated by Sponsor | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo capsule, 20 mg, orally once daily
- Total: Total of all reporting groups
Arm/Group | EGT0001442 | Placebo | Total
Number analyzed (Participants) | 145 | 141 | 286
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (10.94) | 54.7 (10.30) | 55.4 (10.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 91 | 169
  Male | 67 | 50 | 117
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 129 | 125 | 254
  Not Hispanic or Latino | 16 | 16 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 110 | 112 | 222
  More than one race | 31 | 25 | 56
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 29.7 (5.35) | 30.6 (5.41) | 30.1 (5.39)
Baseline HbA1c Category [Count of Participants; unit: Participants]
  < 8.5% | 87 | 100 | 187
  > 8.5% | 58 | 41 | 99

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c at 24 Weeks
Description: Changes from baseline in HbA1c in placebo and treatment group at end of 24 weeks treatment
Time Frame: Baseline and Week 24
Population: Number of subjects with a value at baseline and at the specified visit
Measure: Least Squares Mean (Standard Error); unit: percentage of glycated hemoglobin
Arm/Group | EGT0001442 | Placebo
Number analyzed (Participants) | 140 | 131
percentage of glycated hemoglobin | -0.28 (0.194) | 0.51 (0.200)
Statistical Analysis 1: Comparison: EGT0001442 vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA — The p-value is from a 2-sided t-test for the difference in means of change from baseline. Statistical significant is set at 0.05 level; Based on analysis of covariance, including treatment group, baseline HbA1c, site, age category, gender and race; Difference of LS Means = -0.79, 95% CI 2-sided [-1.06 to -0.53]

2. Secondary Outcome: Changes in Systolic and Diastolic Blood Pressure at Week 24
Description: Changes from baseline in systolic and diastolic blood pressure in placebo and treatment group after 24 weeks of treatment
Time Frame: Baseline and Week 24
Population: Number of subjects with a value at baseline and a the specified visit
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | EGT0001442 | Placebo
Number analyzed (Participants) | 140 | 131
mm Hg
  Systolic blood pressure | -8.62 (1.903) | -3.08 (1.964)
  Diastolic blood pressure | -3.07 (1.223) | -0.40 (1.275)
Statistical Analysis 1: Comparison: EGT0001442 vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Based on analysis of covariance, including treatment group, baseline systolic BP, baseline HbA1c category, site, age category, gender and race; Difference of LS Means = -5.53, 95% CI 2-sided [-8.02 to -3.04]
Statistical Analysis 2: Comparison: EGT0001442 vs Placebo; Test type: Superiority; p = 0.0015, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Based on analysis of covariance, including treatment group, baseline diastolic BP, baseline HbA1c category, site, age category, gender and race; Difference of LS Means = -2.67, 95% CI 2-sided [-4.30 to -1.04]

3. Secondary Outcome: Changes in Body Weight at Week 24
Description: Changes from baseline in body weight in placebo and treatment group after 24 weeks of treatment
Time Frame: Baseline and week 24
Population: Number of subjects with a value at baseline and at the specified visit
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | EGT0001442 | Placebo
Number analyzed (Participants) | 128 | 104
kg | -2.95 (0.555) | -1.22 (0.592)
Statistical Analysis 1: Comparison: EGT0001442 vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Based on analysis of covariance, including treatment group, baseline weight, baseline HbA1c category, site, age category, gender and race; Difference of LS Means = -1.72, 95% CI 2-sided [-2.52 to -0.93]

4. Secondary Outcome: Change From Baseline in HbA1c Over 96 Weeks Time
Description: Change from baseline in HbA1c level over 96 weeks in placebo and treatment group. The treatment group was treated with EGT0001442 for 24 weeks.
Time Frame: Baseline and up to 96 weeks
Population: Number of subjects with a value at baseline and at the specified visit
Measure: Least Squares Mean (Standard Error); unit: percentage glycated hemoglobin
Arm/Group | EGT0001442 | Placebo
Number analyzed (Participants) | 136 | 128
percentage glycated hemoglobin
  Week 2 | -0.10 (0.083) | 0.22 (0.084)
  Week 6 | -0.11 (0.137) | 0.49 (0.141)
  Week 12 | -0.19 (0.180) | 0.53 (0.186)
  Week 18 | -0.28 (0.195) | 0.43 (0.201)
  Week 24 | -0.28 (0.194) | 0.51 (0.200)
  Week 36 | -0.52 (0.202) | 0.42 (0.209)
  Week 48 | -0.45 (0.215) | 0.54 (0.222)
  Week 60 | -0.57 (0.219) | 0.41 (0.226)
  Week 72 | -0.43 (0.213) | 0.50 (0.220)
  Week 84 | -0.60 (0.218) | 0.38 (0.225)
  Week 96 | -0.48 (0.215) | 0.54 (0.222)
Statistical Analysis 1: Comparison: EGT0001442 vs Placebo; Change from baseline in HbA1c (%) at Week 2; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Based on analysis of covariance, including treatment group, baseline HbA1c, site, age category, gender and race; Difference of LS Means = -0.32, 95% CI 2-sided [-0.42 to -0.21]
Statistical Analysis 2: Comparison: EGT0001442 vs Placebo; Change from baseline in HbA1c (%) at Week 6; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Based on analysis of covariance, including treatment group, baseline HbA1c, site, age category, gender and race; Difference of LS Means = -0.59, 95% CI 2-sided [-0.78 to -0.41]
Statistical Analysis 3: Comparison: EGT0001442 vs Placebo; Change from baseline in HbA1c (%) at Week 12; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Based on analysis of covariance, including treatment group, baseline HbA1c, site, age category, gender and race; Difference of LS Means = -0.72, 95% CI 2-sided [-0.96 to -0.48]
Statistical Analysis 4: Comparison: EGT0001442 vs Placebo; Change from baseline in HbA1c (%) at Week 18; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Based on analysis of covariance, including treatment group, baseline HbA1c, site, age category, gender and race; Difference of LS Means = -0.71, 95% CI 2-sided [-0.97 to -0.44]
Statistical Analysis 5: Comparison: EGT0001442 vs Placebo; Change from baseline in HbA1c (%) at Week 24; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Based on analysis of covariance, including treatment group, baseline HbA1c, site, age category, gender and race; Difference of LS Means = -0.79, 95% CI 2-sided [-1.06 to -0.53]
Statistical Analysis 6: Comparison: EGT0001442 vs Placebo; Change from baseline in HbA1c (%) at Week 36; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Based on analysis of covariance, including treatment group, baseline HbA1c, site, age category, gender and race; Difference of LS Means = -0.93, 95% CI 2-sided [-1.21 to -0.66]
Statistical Analysis 7: Comparison: EGT0001442 vs Placebo; Change from baseline in HbA1c (%) at Week 48; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Based on analysis of covariance, including treatment group, baseline HbA1c, site, age category, gender and race; Difference of LS Means = -0.99, 95% CI 2-sided [-1.28 to -0.70]
Statistical Analysis 8: Comparison: EGT0001442 vs Placebo; Change from baseline in HbA1c (%) at Week 60; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Based on analysis of covariance, including treatment group, baseline HbA1c, site, age category, gender and race; Difference of LS Means = -0.98, 95% CI 2-sided [-1.27 to -0.68]
Statistical Analysis 9: Comparison: EGT0001442 vs Placebo; Change from baseline in HbA1c (%) at Week 72; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Based on analysis of covariance, including treatment group, baseline HbA1c, site, age category, gender and race; Difference of LS Means = -0.93, 95% CI 2-sided [-1.22 to -0.64]
Statistical Analysis 10: Comparison: EGT0001442 vs Placebo; Change from baseline in HbA1c (%) at Week 84; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Based on analysis of covariance, including treatment group, baseline HbA1c, site, age category, gender and race; Difference of LS Means = -0.98, 95% CI 2-sided [-1.27 to -0.69]
Statistical Analysis 11: Comparison: EGT0001442 vs Placebo; Change from baseline in HbA1c (%) at Week 96; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Based on analysis of covariance, including treatment group, baseline HbA1c, site, age category, gender and race; Difference of LS Means = -1.02, 95% CI 2-sided [-1.31 to -0.73]

5. Secondary Outcome: Change From Baseline Over Time in Fasting Plasma Glucose (FPG)
Description: Changes from baseline in FPG in placebo and treatment group over 24 weeks of treatment
Time Frame: 24 weeks
Population: Only included number of subjects with a value at baseline and at the specified visit
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | EGT0001442 | Placebo
Number analyzed (Participants) | 145 | 138
mmol/L
  Week 2: number analyzed (Participants) | 138 | 127
  Week 2 | -1.39 (0.407) | 0.85 (0.422)
  Week 6: number analyzed (Participants) | 139 | 131
  Week 6 | -1.23 (0.482) | 1.22 (0.499)
  Week 12: number analyzed (Participants) | 140 | 131
  Week 12 | -1.75 (0.489) | 0.67 (0.507)
  Week 18: number analyzed (Participants) | 140 | 131
  Week 18 | -1.87 (0.451) | 0.83 (0.467)
  Week 24: number analyzed (Participants) | 140 | 131
  Week 24 | -1.74 (0.462) | 0.89 (0.478)
Statistical Analysis 1: Comparison: EGT0001442 vs Placebo; Difference of mean-adjusted change from baseline in FPG (mmol/L) at Week 2, between EGT0001442 and Placebo group; Test type: Superiority; p < 0.0001, ANCOVA — The p-value is from a two-sided t-test for the difference in means of change from baseline; Based on analysis of covariance, including treatment group, baseline FPG, baseline HbA1c category, site, age category, gender and race; Difference of LS Means = -2.24, 95% CI 2-sided [-2.79 to -1.70]
Statistical Analysis 2: Comparison: EGT0001442 vs Placebo; Difference of mean-adjusted change from baseline in FPG (mmol/L) at Week 6, between EGT0001442 and Placebo group; Test type: Superiority; p < 0.0001, ANCOVA — The p-value is from a two-sided t-test for the difference in means of change from baseline; [statistical method as in outcome 5, analysis 1]; Difference of LS Means = -2.45, 95% CI 2-sided [-3.09 to -1.81]
Statistical Analysis 3: Comparison: EGT0001442 vs Placebo; Difference of mean-adjusted change from baseline in FPG (mmol/L) at Week 12, between EGT0001442 and Placebo group; Test type: Superiority; p < 0.0001, ANCOVA — The p-value is from a two-sided t-test for the difference in means of change from baseline; [statistical method as in outcome 5, analysis 1]; Difference of LS Means = -2.42, 95% CI 2-sided [-3.06 to -1.77]
Statistical Analysis 4: Comparison: EGT0001442 vs Placebo; Difference of mean-adjusted change from baseline in FPG (mmol/L) at Week 18, between EGT0001442 and Placebo group; Test type: Superiority; p < 0.0001, ANCOVA — The p-value is from a two-sided t-test for the difference in means of change from baseline; [statistical method as in outcome 5, analysis 1]; Difference of LS Means = -2.71, 95% CI 2-sided [-3.30 to -2.11]
Statistical Analysis 5: Comparison: EGT0001442 vs Placebo; Difference of mean-adjusted change from baseline in FPG (mmol/L) at Week 24, between EGT0001442 and Placebo group; Test type: Superiority; p < 0.0001, ANCOVA — The p-value is from a two-sided t-test for the difference in means of change from baseline; [statistical method as in outcome 5, analysis 1]; Difference of LS Means = -2.63, 95% CI 2-sided [-3.24 to -2.02]

6. Secondary Outcome: Percentage of Subjects Achieving HbA1c <7%
Description: The number and percentage of subjects achieving HbA1c response levels <7% for the FAS using LOCF is reported
Time Frame: Baseline and up to 96 weeks
Population: Only included number of subjects with a value at baseline and at the specified visit
Measure: Count of Participants; unit: Participants
Arm/Group | EGT0001442 | Placebo
Number analyzed (Participants) | 145 | 138
Participants
  Week 2: number analyzed (Participants) | 136 | 128
  Week 2 | 14 | 13
  Week 6: number analyzed (Participants) | 139 | 131
  Week 6 | 22 | 15
  Week 12: number analyzed (Participants) | 140 | 131
  Week 12 | 27 | 17
  Week 18: number analyzed (Participants) | 140 | 131
  Week 18 | 29 | 14
  Week 24: number analyzed (Participants) | 140 | 131
  Week 24 | 33 | 14
  Week 36: number analyzed (Participants) | 140 | 131
  Week 36 | 35 | 14
  Week 48: number analyzed (Participants) | 140 | 131
  Week 48 | 41 | 20
  Week 60: number analyzed (Participants) | 140 | 131
  Week 60 | 39 | 18
  Week 72: number analyzed (Participants) | 140 | 131
  Week 72 | 39 | 17
  Week 84: number analyzed (Participants) | 140 | 131
  Week 84 | 43 | 16
  Week 96: number analyzed (Participants) | 140 | 131
  Week 96 | 44 | 14

ADVERSE EVENTS:
Time Frame: The adverse event data were collected from Week 0 (Visit 3) up to Week 97 (Visit 15, 1 week follow-up after completion of study).
Arm/Group | EGT0001442 | Placebo
All-Cause Mortality (participants affected / at risk) | 1/145 | 0/141
Serious Adverse Events (participants affected / at risk) | 3/145 | 12/141
Other Adverse Events (participants affected / at risk) | 50/145 | 62/141
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EGT0001442 (N=145) | Placebo (N=141)
Cardiac arrest (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Hypertensive crisis (Cardiac disorders) | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 2 | 0
Diverticulitis (Gastrointestinal disorders) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Spinal column stenosis (Nervous system disorders) | 0 | 1
Peripheral nerve lesion (Nervous system disorders) | 0 | 1
Acute polyneuropathy (Nervous system disorders) | 0 | 1
Lumbar spinal stenosis (Nervous system disorders) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EGT0001442 (N=145) | Placebo (N=141)
Hypoglycemia (Metabolism and nutrition disorders) | 24 | 24
Dyslipidaemia (Metabolism and nutrition disorders) | 5 | 8
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 5 | 8
Urinary Tract Infection (Infections and infestations) | 17 | 28
Headache (Nervous system disorders) | 7 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI is not allowed to publish trial results.

DOCUMENTS (2):
  • Study Protocol (2011-02-02): https://cdn.clinicaltrials.gov/large-docs/44/NCT01377844/Prot_000.pdf
  • Statistical Analysis Plan (2011-11-22): https://cdn.clinicaltrials.gov/large-docs/44/NCT01377844/SAP_001.pdf